CLINICAL TRIAL: NCT05332873
Title: Safety and Efficacy of the Rivet Pulmonary-to-Venous Shunt (PVS) Therapy in Patients With Group 2 Pulmonary Hypertension (PH) Due to Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Rivet PVS Therapy in Group 2 PH-HFpEF Canada
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Commercial decision
Sponsor: NXT Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-A-21-0001-CAN
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Rivet Shunt Therapy (Experimental)
  Interventions: Device: Rivet Shunt

INTERVENTIONS:
Device: Rivet Shunt — The Rivet Shunt device will be implanted via a percutaneous, transcatheter approach

SUMMARY:
This clinical investigation is a prospective, multicenter, non-randomized, open-label, Early Feasibility Study to evaluate the safety, performance, and initial clinical efficacy of the Rivet PVS therapy in patients with symptomatic pulmonary hypertension.

ELIGIBILITY:
Select Inclusion Criteria:

* Age ≥ 18 years
* Prior diagnosis of Group 2 PH due to HFpEF, with at least one of the following resting hemodynamic criteria confirmed in the past year by right heart catheterization

  1. mPAP > 20 mmHg at rest
  2. mPAP/CO slope > 3 mmHg/L/min with exercise
* Confirmation of the following hemodynamic criteria during supine exercise: PCWP ≥ 25 mmHg, or PCWP/CO slope > 2 mmHg/L/min
* Chronic symptomatic heart failure documented by the following:

  1. NYHA HF Class II with history > II, or Class III, or ambulatory Class IV
  2. ≥ 1 HF hospitalization, or healthcare facility with IV diuretics or intensification of oral diuresis for HF within 12 months, or NT-pro BNP value > 400 pg/mL in normal sinus rhythm or > 750 pg/mL in atrial fibrillation in past 6 months
* Ongoing stable guideline directed medical therapy (GDMT) for HF and medically optimized per treating cardiologist according to current ACCF/AHA guidelines that is expected to be maintained without change for 1 month (excluding diuretic dosage changes for HF optimization within 30 days of the Index Procedure)
* 6MWD ≥ 100 m

Select Exclusion Criteria:

* Any therapeutic intracardiac intervention within the last 30 days
* PH Group 1, 3, 4 or 5
* Mean RAP >16 mmHg by RHC at rest on room air
* Right ventricular dysfunction, defined as one or more of the following

  1. Greater than moderate RV dysfunction as assessed by TTE and/or MRI
  2. RV FAC < 35%
  3. TAPSE < 14 mm via TTE
  4. RV size severely enlarged compared to LV size as estimated by TTE and/or MRI
* Severe tricuspid valve regurgitation
* Peak systolic pulmonary arterial pressure > 80 mmHg by RHC at rest while awake
* Mean pulmonary arterial pressure > 50 mmHg by RHC at rest while awake
* PVR > 6 Wood units at rest while awake on room air
* Left ventricular ejection fraction < 50%
* Severe heart failure, defined as one or more of the following:

  1. ACC/AHA/ESC Stage D heart failure, non-ambulatory NYHA Class IV HF
  2. If BMI < 30, Cardiac Index < 2.0 L/min/m2
  3. If BMI ≥ 30, Cardiac Index < 1.8 L/min/m2
  4. Requires continuous intravenous inotropic infusion
  5. Requires mechanical circulatory support
  6. Currently on the cardiac transplant waiting list
* Chronic renal dysfunction defined as: eGFR < 35 mL/min/1.73 m2 by the CKD-Epi equation
* Chronic pulmonary disease defined as one or more of the following:

  1. Requires continuous home oxygen therapy
  2. Recent hospitalization for exacerbation within 12 months prior to screening
  3. FEV1 < 50% predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events | 1 month
  Composite of major adverse cardiac, cerebrovascular, or renal events (MACCRE) and re-intervention for study device related complications at implantation procedure (Day 0) and up to 1-month post-procedure (Day 30)
Rate of Technical Success of the Rivet Shunt Implantation Procedure | At time of procedure
  Study device is implanted as intended and confirmation of a patent pulmonary-to-venous shunt between the RPA and SVC by qualitative assessment via angiography and/or echocardiography at implantation procedure.

SECONDARY OUTCOMES:
Adverse Events through 12 months | 12 months
  Composite of MACCRE and re-intervention for study device related complications (as described above), progression of PH and/or HF disease, and all-cause mortality to 12 months post-procedure
Change in Hemodynamics at 12 months - PCWP | 12 Months
  Change in exercise pulmonary capillary wedge pressure (PCWP) from baseline
Change in Kansas City Cardiomyopathy Questionnaire | 12 months
  Change in KCCQ score between baseline and 12 months.
Change in RV Chamber Size at 12 months - Diameter | 12 months
  Change in RV Chamber Size (Diameter) assessed by a core lab between baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No